CLINICAL TRIAL: NCT07386015
Title: FREEZE-Path Cohort: Etiology-Phenotype-Outcome Pathway Study on Freezing of Gait (FOG)
Brief Title: Etiology-Phenotype-Outcome Pathway Study on Freezing of Gait (FOG)
Status: Not yet recruiting | Type: Observational
Sponsor: Tianjin Huanhu Hospital (Other)
Responsible Party: Principal Investigator, Peipei Liu, Principal Investigator, Tianjin Huanhu Hospital
Other Study IDs: (Jin Huan) 2025-297
Record Dates: First submitted 2025-12-24; First posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Freezing of Gait; Parkinson's Disease; Parkinsonism; Vascular Parkinsonism; Idiopathic Normal Pressure Hydrocephalus (INPH)
Keywords: Freezing of Gait; Parkinson's Disease; parkinsonism
MeSH Terms: conditions — Parkinson Disease; Parkinsonian Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 36 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- FOG Group: This cohort includes participants with freezing of gait present at baseline. Participants may have Parkinson's disease or other neurological conditions associated with freezing of gait. All participants receive standard clinical care as determined by their treating physicians. No experimental treatments or study-specific interventions are assigned as part of this observational registry.
  Interventions: Other: Observational Data Collection
- High-Risk Group: This cohort includes participants with gait or balance impairment who have not developed freezing of gait at baseline but are considered at high risk for future freezing of gait. Participants may have Parkinson's disease or related neurological disorders. All participants receive standard clinical care, and no experimental treatments or study-specific interventions are provided as part of this observational registry.
  Interventions: Other: Observational Data Collection

INTERVENTIONS:
Other: Observational Data Collection — This is an observational patient registry. No experimental drugs, devices, or procedures are assigned as part of the study. All participants receive standard medical care, and data are collected during routine clinical visits and follow-up assessments.

SUMMARY:
This study is a prospective, multicenter, observational cohort (patient registry) designed to better understand freezing of gait (FOG), a disabling walking problem that can occur in Parkinson's disease and other related neurological conditions.The purpose of this registry is to collect long-term clinical information from patients with freezing of gait or gait and balance problems, and to explore how different causes of FOG are related to symptoms, walking patterns, falls, disease progression, and outcomes over time. The study will include participants with Parkinson's disease and other conditions associated with freezing of gait.Participants will receive standard medical care as determined by their treating physicians. No experimental drugs or study-related treatments will be assigned as part of this registry. Clinical information will be collected during routine visits and follow-up assessments, including questionnaires, walking and balance evaluations, video recordings, and other commonly used clinical tests.The information collected in this study may help improve the understanding of freezing of gait, support better risk assessment for falls, and guide future research and clinical management strategies for patients with gait and balance disorders.

DETAILED DESCRIPTION:
Freezing of gait (FOG) is a common and disabling gait disturbance characterized by a transient inability to initiate or maintain effective stepping. It is most frequently observed in Parkinson's disease but can also occur in other parkinsonian syndromes and neurological conditions associated with gait and balance dysfunction. Freezing of gait is associated with falls, loss of independence, reduced quality of life, and increased caregiver burden, yet its underlying mechanisms, clinical heterogeneity, and long-term trajectories remain incompletely understood.

This study is a prospective, multicenter, observational patient registry designed to systematically collect longitudinal clinical data from adults with freezing of gait, gait and balance impairment, or those at high risk for developing freezing of gait. Participants will be recruited from neurology and related specialty clinics at participating centers and followed over time as part of routine clinical care.

The registry will collect a broad range of clinical information, including but not limited to:

Demographic and clinical characteristics; Freezing of gait severity and related symptoms; Objective gait parameters and balance performance assessed using standardized gait tasks; Motor symptom severity and functional status; Falls and fall-related outcomes; Health-related quality of life and other patient-reported outcomes. Clinical assessments will be performed at baseline and during scheduled follow-up visits over a planned follow-up period of up to 36 months. Data collection may include questionnaires, clinician-rated scales, objective gait and balance assessments, and video-based evaluations, depending on local clinical practice and participant capability.

This registry is non-interventional. All diagnostic and therapeutic decisions, including medication adjustments and rehabilitative interventions, will be made solely by the treating physicians according to standard clinical practice. The study does not mandate any experimental drugs, devices, or procedures.

The primary objectives of this registry are to:

Characterize the longitudinal course and clinical variability of freezing of gait; Examine associations between freezing of gait, gait and balance impairment, falls, and clinical outcomes; Identify potential clinical phenotypes and risk factors associated with worsening gait dysfunction and adverse outcomes.

The findings from this registry are intended to support hypothesis generation, improve clinical risk assessment, and provide a foundation for the development of future mechanistic studies and interventional trials targeting freezing of gait and related gait disorders.

ELIGIBILITY:
Inclusion Criteria:

1. Age 30-85 years
2. Presence of freezing of gait or non-freezing gait or balance impairment
3. Diagnosis of Parkinson's disease or related parkinsonian disorders according to established international criteria (including PD, PSP, MSA, DLB, CBD, vascular parkinsonism, or idiopathic normal pressure hydrocephalus)
4. Ability to complete gait and balance assessment tasks independently or with assistance
5. Ability and willingness to provide written informed consent

Exclusion Criteria:

1. Severe dementia (Mini-Mental State Examination score < 10)
2. Severe psychiatric disorders interfering with study participation
3. Severe cardiopulmonary, musculoskeletal, or other medical conditions significantly affecting gait safety
4. Stroke, fracture, or other major medical events within the past 3 months
5. Inability to comply with follow-up procedures
6. Refusal of video or speech data collection

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population includes adults aged 30 to 85 years with freezing of gait or gait and balance impairment. Participants are diagnosed with Parkinson's disease or other parkinsonian or related neurological disorders associated with freezing of gait, including but not limited to parkinsonian syndromes and other causes of gait dysfunction.
  Both participants with established freezing of gait and participants at high risk for developing freezing of gait are included. All participants are recruited from neurology and related specialty clinics at participating centers and are followed longitudinally as part of a prospective observational patient registry.
Sampling Method: Non-Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2026-02-10 (Estimated); Primary Completion 2029-12-31 (Estimated); Study Completion 2030-11-30 (Estimated)

PRIMARY OUTCOMES:
Change in Freezing of Gait Severity Measured by the New Freezing of Gait Questionnaire (NFOG-Q) | Baseline to 36 months
  The New Freezing of Gait Questionnaire (NFOG-Q) is a patient-reported outcome measure assessing the severity and impact of freezing of gait in Parkinson's disease.
  The total score ranges from 0 to 28, with higher scores indicating more severe freezing of gait.
  The primary outcome is the change in NFOG-Q total score from baseline to 36 months.

SECONDARY OUTCOMES:
Time to First Freezing of Gait Event | Baseline to 36 months
  Time from baseline to the first occurrence of freezing of gait in participants without freezing of gait at baseline.
Frequency of Falls | Baseline to 36 months
  Number of falls reported during follow-up, collected through clinical visits and follow-up assessments.
Change in Health-Related Quality of Life Measured by the Parkinson's Disease Questionnaire-39 (PDQ-39) | Baseline to 36 months
  Health-related quality of life will be assessed using the Parkinson's Disease Questionnaire-39 (PDQ-39), a validated patient-reported outcome measure for individuals with Parkinson's disease.
  The PDQ-39 Summary Index score ranges from 0 to 100, with higher scores indicating worse health-related quality of life.
  The outcome is defined as the change in PDQ-39 Summary Index score from baseline to 36 months.
Change in Gait Speed | Baseline to 36 months
  Gait speed will be measured during standardized gait tasks using an objective gait assessment system.
  The outcome is defined as the change in gait speed (meters per second, m/s) from baseline to 36 months, with higher values indicating better gait performance.
Change in Stride Length | Baseline to 36 months
  Stride length will be assessed during standardized gait tasks using an objective gait assessment system.
  The outcome is defined as the change in stride length (meters, m) from baseline to 36 months, with higher values indicating better gait performance.
Change in Gait Variability | Baseline to 36 months
  Gait variability will be quantified during standardized gait tasks using an objective gait assessment system.
  Gait variability will be expressed as the coefficient of variation (%) of stride length.
  The outcome is defined as the change in gait variability from baseline to 36 months, with lower values indicating better gait stability.
Change in Balance Performance Measured by the Mini-Balance Evaluation Systems Test (Mini-BESTest) | Baseline to 36 months
  Balance performance will be assessed using the Mini-Balance Evaluation Systems Test (Mini-BESTest), a validated clinical scale for evaluating dynamic balance in patients with Parkinson's disease.
  The Mini-BESTest total score ranges from 0 to 28, with higher scores indicating better balance performance.
  The outcome is defined as the change in Mini-BESTest total score from baseline to 36 months.
Changes in functional brain network connectivity assessed by resting-state functional MRI (fMRI) | Baseline to 36 months.
  This outcome evaluates longitudinal changes in fMRI-derived functional connectivity within and between frontal cortical regions, basal ganglia, and brainstem locomotor control areas. The objective is to construct an integrated "brain network-clinical phenotype-FOG outcome" framework, enabling identification of neural network signatures specifically associated with freezing of gait and its progression.

CONTACTS AND LOCATIONS:
Overall Officials: Peipei Liu, MD, Principal Investigator — Tianjin Huanhu Hospital
Locations (1):
- Tianjin Huanhu Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] 1.Talia H, Yael B, Michal B, et al.: A meta-analysis identifies factors predicting the future development of freezing of gait in parkinson's disease[J]. NPJ Parkinsons Dis 2023, 9.10.1038/s41531-023-00600-2. 2.Richard C, Meg E M, Frederico P-F, et al.: Prevention of falls in parkinson's disease: Guidelines and gaps[J]. Mov Disord Clin Pract 2023, 10.10.1002/mdc3.13860. 3.Seira T, Yuta K, Takanori K, et al.: New insights into freezing of gait in parkinson's disease from spectral dynamic causal modeling[J]. Mov Disord 2024, 39.10.1002/mds.29988. 4.Giladi N, Nieuwboer A. Understanding and treating freezing of gait in Parkinson's disease: a review of current concepts and future directions. Lancet Neurology. 2008;7(8):720-730. 5.Kelvin L C, Prabesh K, Miriam vEB, et al.: Cholinergic system changes in dopa-unresponsive freezing of gait in parkinson's disease[J]. Mov Disord 2025, 40.10.1002/mds.30196.

DOCUMENTS (2):
  • Study Protocol (2025-10-20): https://cdn.clinicaltrials.gov/large-docs/15/NCT07386015/Prot_000.pdf
  • Informed Consent Form (2025-10-20): https://cdn.clinicaltrials.gov/large-docs/15/NCT07386015/ICF_001.pdf